CLINICAL TRIAL: NCT07404033
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase Ⅰb Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Different Concentrations of ZYG24002 Lotion in Adult Patients With Mild to Moderate Seborrheic Dermatitis
Brief Title: ZYG24002 Lotion to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy in Adult Patients With Mild to Moderate Seborrheic Dermatitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sinomune Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYG-24002-Ⅰ-01-2025-02
Record Dates: First submitted 2026-01-25; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Seborrheic Dermatitis
Keywords: seborrheic dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZYG24002 0.5%， BID (Experimental): Participants apply 0.5% concentration or placebo ZYG24002 Lotion twice daily (BID) for a consecutive period of 28 days.
  Interventions: Drug: ZYG24002 0.5%; Drug: ZYG24002 Placebo
- ZYG24002 0.75% ,BID (Experimental): Participants apply 0.75% concentration or placebo ZYG24002 Lotion twice daily (BID) for a consecutive period of 28 days.
  Interventions: Drug: ZYG24002 0.75%; Drug: ZYG24002 Placebo
- ZYG24002 1%, BID (Experimental): Participants apply 1% concentration or placebo ZYG24002 Lotion twice daily (BID) for a consecutive period of 28 days.
  Interventions: Drug: ZYG24002 1%; Drug: ZYG24002 Placebo
- ZYG24002 1%, QD (Experimental): Participants apply 1% concentration or placebo ZYG24002 Lotion once daily (QD) for a consecutive period of 28 days.
  Interventions: Drug: ZYG24002 1%; Drug: ZYG24002 Placebo

INTERVENTIONS:
Drug: ZYG24002 0.5% — 0.5% concentration of ZYG24002
  Arms: ZYG24002 0.5%， BID
Drug: ZYG24002 0.75% — 0.75% concentration of ZYG24002
  Arms: ZYG24002 0.75% ,BID
Drug: ZYG24002 1% — 1% concentration of ZYG24002
  Arms: ZYG24002 1%, BID; ZYG24002 1%, QD
Drug: ZYG24002 Placebo — 0% concentration of ZYG24002

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase Ib clinical trial conducted in adult patients with mild to moderate seborrheic dermatitis (IGA-SD score of 2-3 points). The study aims to evaluate the safety, tolerability, and steady-state pharmacokinetic (PK) profiles of three concentrations (0.5%, 0.75%, and 1.0%) of ZYG24002 Lotion following continuous topical application once daily (QD) or twice daily (BID) for 28 days, and to conduct a preliminary exploration of the drug's efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 (inclusive) to 65 (inclusive) years, of either sex. Male subjects must have no childbearing potential or agree to adopt contraceptive measures until 3 months after the end of the study; female subjects of childbearing potential must be non-pregnant and non-lactating, and adopt reliable contraceptive measures during the study period and within 3 months after the last dose.
2. Diagnosed with seborrheic dermatitis by a dermatologist (diagnostic criteria refer to the Expert Consensus on Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment of Seborrheic Dermatitis (2024 Edition) and the 2015 Asian Consensus on Seborrheic Dermatitis), with a disease duration of ≥ 3 months; baseline Investigator's Global Assessment for Seborrheic Dermatitis (IGA-SD) score (0-4 point scale) of 2 (mild) or 3 (moderate); at baseline, the overall scores for erythema and scaling are at least mild severity (score 1) respectively. The involved body surface area (BSA%) is ≤ 10%, and skin lesions are distributed in at least two anatomical sites such as the scalp, face, and trunk.
3. No obvious signs of infection at the test site (e.g., pustules, crusts caused by bacterial infection). The subject is in good general skin condition at enrollment, with no other active skin lesions that may interfere with the clinical assessment.
4. Has not participated in any other clinical trials or used any investigational drugs within the past 3 months.
5. Study participants provide informed consent to participate in this study, sign the informed consent form (ICF), are able to understand the study requirements, and are willing to complete all scheduled visits and examinations in accordance with the investigator's instructions.

Exclusion Criteria:

1. Severe active seborrheic dermatitis: IGA-SD score of 4 points or extensive skin lesions (BSA > 10%), accompanied by obvious exudation and infection, requiring systemic therapy. Participants whose disease activity is deemed unsuitable for study enrollment by the investigator (including but not limited to situations where 4 weeks of placebo-only treatment may lead to unacceptable disease progression).
2. Comorbidities of other skin diseases that may interfere with study assessments, such as psoriasis, severe acne, rosacea, atopic dermatitis, etc., which would confound the observation of seborrheic dermatitis lesions.
3. Administration of systemic glucocorticoids, systemic retinoids, immunosuppressants, oral/intravenous antifungals, phototherapy, PDE-4 inhibitors, or JAK inhibitors within 4 weeks; topical glucocorticoids, calcineurin inhibitors, PDE-4 inhibitors, antifungals, retinoids, keratolytics, selenium/tar-containing preparations on the study area within 2 weeks; any biologic agents within 6 months; or potent CYP3A4 inhibitors/inducers within 4 weeks.
4. Receipt of physical or chemical cosmetic treatments on the head and face within the past month (e.g., intense pulsed light, glycolic acid peels), resulting in temporary skin barrier dysfunction that has not yet recovered to normal.
5. A history of known severe hypersensitivity or severe adverse reactions to ZYG24002 or its excipients.
6. Comorbidities of other skin diseases that may increase the systemic absorption of ZYG24002, such as Netherton syndrome or erythroderma.
7. Current use of immunosuppressants or diagnosis of immune deficiency.
8. A history of malignancy within 5 years prior to screening or at screening.
9. Poorly controlled chronic diseases, including but not limited to endocrine disorders (e.g., diabetes mellitus with significantly elevated fasting blood glucose and obvious clinical symptoms, hyperthyroidism); a history of severe cardiovascular and cerebrovascular diseases (e.g., myocardial infarction, stroke); active peptic ulcers or chronic inflammatory bowel disease, etc.
10. Abnormal liver function: ALT or AST > 2 × upper limit of normal (ULN), or total bilirubin > 1.5 × ULN at screening; abnormal renal function: serum creatinine > 1.5 × ULN; or other clinically significant abnormal laboratory findings that are deemed unsuitable for enrollment by the investigator.
11. Human immunodeficiency virus (HIV) infection; active hepatitis C virus (HCV) infection (anti-HCV positive); active hepatitis B virus (HBV) infection (HBV-DNA > 2000 IU/mL or 10⁴ CPs/mL); or positive treponema pallidum antibody with evidence of active infection.
12. Diagnosis of psychiatric or neurological disorders that may affect compliance or increase study-related risks.
13. Pregnancy, lactation, or planned pregnancy; female subjects of childbearing potential who have not initiated reliable contraceptive measures at least 30 days prior to the first dose and who cannot commit to maintaining such measures for 3 months after the last dose.
14. Diagnosis of alcohol or addictive substance dependence within the past 12 months, or other conditions that the investigator believes may compromise study compliance.
15. Any other conditions that the investigator deems may interfere with study results or pose an unacceptable safety risk to the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rates of Serious Adverse Events (SAE) during the trial period | Through study completion, an average of 1 year
  Safety assessment will include the types and incidence rates of all serious adverse events (SAE) occurring during the study period; and the causal relationship between SAE and the study drug (assessed using a five-level evaluation method: Definite, Probable, Possible, Unlikely, Unrelated).
The incidence rate of adverse events (AE) occurring during the treatment period with severity grade ≥ 3 | Through study completion, an average of 1 year
  Calculate the incidence rate of adverse events (AE) occurring during the treatment period with severity grade ≥ 3 (per CTCAE V5.0 criteria) ; record the specific types, severity, and causal relationship with the study drug of the aforementioned treatment-emergent adverse events (TEAE).
The incidence rate of adverse events (AE) occurring during the treatment period resulting in treatment discontinuation | Through study completion, an average of 1 year
  Calculate the incidence rate of adverse events (AE) occurring during the treatment period with resulting in treatment discontinuation; record the specific types, severity, and causal relationship with the study drug of the aforementioned treatment-emergent adverse events (TEAE).
Local Tolerability (LT) Indicator: the proportion of study participants with local cutaneous reactions of severity grade ≥ 2 during the study period | Through study completion, an average of 1 year
  Calculate the proportion of study participants with local cutaneous reactions (including stinging sensation, burning sensation, pruritus, erythema, and edema/papules) of severity grade ≥ 2 during the study period
Local Tolerability (LT) Indicator: the proportion of study participants with treatment interruption or discontinuation due to local tolerability adverse reactions | Through study completion, an average of 1 year
  Record the proportion of study participants with treatment interruption or discontinuation due to local tolerability adverse reactions, as well as the occurrence frequency, types, and trends of change of the aforementioned local tolerability reactions.
Supportive Safety Endpoints - The incidence rate of Adverse Events (AE) (including Grade 1-2) | Through study completion, an average of 1 year
  Record the types, incidence rates, severity, and drug-relatedness of all adverse events (AE) (including Grade 1-2) occurring during the treatment period (Day 1 - Day 35 ± 2)
Supportive Safety Endpoints - the incidence rate of abnormalities in vital signs (blood pressure [BP], heart rate [HR], body temperature [BT]) | Through study completion, an average of 1 year
  Calculate the incidence rate of abnormalities in vital signs (blood pressure [BP], heart rate [HR], body temperature [BT]); Record the changes in vital signs (blood pressure [BP], heart rate [HR], body temperature [BT]) and their clinical significance among study participants in each dose group during the treatment and follow-up periods
Supportive Safety Endpoints - The incidence rate of abnormalities in laboratory test indicators (including blood routine, blood biochemistry, urine routine) | Through study completion, an average of 1 year
  Calculate the incidence rate and severity of abnormalities in laboratory test indicators (including blood routine, blood biochemistry, urine routine) among study participants in each dose group during the treatment and follow-up periods
Supportive Safety Endpoints - The incidence rate of abnormalities in electrocardiogram (ECG) examinations | Through study completion, an average of 1 year
  Calculate the incidence rate of abnormalities in electrocardiogram (ECG) examinations and their clinical significance among study participants in each dose group during the treatment and follow-up periods

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Up to 24 hours after first dose
  Peak concentration (Cmax) after a single dose
Time to peak concentration (Tmax) | Up to 24 hours after first dose
  Time to peak concentration (Tmax) after a single dose
Single-dose exposure (Area Under the Curve from 0 to τ, AUC0-τ, τ=24 h for QD, τ=12 h for BID) | Up to 24 hours after first dose
  Single-dose exposure (Area Under the Curve from 0 to τ, AUC0-τ, τ=24 h for QD, τ=12 h for BID)
Steady-state peak concentration (Cmax,ss) | Day 29
  Steady-state peak concentration (Cmax,ss)
Steady-state trough concentration (Cmin,ss) | Day 29
  Steady-state trough concentration (Cmin,ss)
Accumulation ratio (Rac): The ratio of steady-state Cmax,ss to single-dose Cmax | Day 29
  Accumulation ratio (Rac): The ratio of steady-state Cmax,ss to single-dose Cmax
Accumulation ratio (Rac): the ratio of steady-state AUC to single-dose AUC | Day 29
  Accumulation ratio (Rac): the ratio of steady-state AUC to single-dose AUC
IGA-SD Treatment Success Rate after treatment on Day 15±1 | Day 15
  Defined as the proportion of study participants whose Investigator's Global Assessment for Seborrheic Dermatitis (IGA-SD, 0-4 point scale) score of the target area reaches 0 (Clearance) or 1 (Near Clearance) after treatment on Day 15±1 , with an improvement of ≥ 2 grades from baseline.
IGA-SD Treatment Success Rate after treatment on Day 29 | Day 29
  Defined as the proportion of study participants whose Investigator's Global Assessment for Seborrheic Dermatitis (IGA-SD, 0-4 point scale) score of the target area reaches 0 (Clearance) or 1 (Near Clearance) after treatment on Day 29, with an improvement of ≥ 2 grades from baseline.
Change in Total Erythema Score on Day 15±1 | Day 15
  The change in total erythema score (0-3 point scale) on Day 15±1 compared with baseline
Change in Total Erythema Score on Day 29 | Day 29
  The change in total erythema score (0-3 point scale) on Day 29 compared with baseline
Change in Total Scaling Score on Day 15±1 | Day 15
  The change in total scaling score (0-3 point scale) on Day 15±1 compared with baseline
Change in Total Scaling Score on Day 29 | Day 29
  The change in total scaling score (0-3 point scale) on Day 29 compared with baseline
Change in Worst Itch Intensity (WI-NRS) on Day 15±1 | Day 15
  The change in Worst Itch Intensity (WI-NRS, 0-10 point scale) on Day 15±1 compared with baseline
Change in Worst Itch Intensity (WI-NRS) on Day 29 | Day 29
  The change in Worst Itch Intensity (WI-NRS, 0-10 point scale) on Day 29 compared with baseline
Change in DLQI Score | Day 29
  The change in Dermatology Life Quality Index (DLQI) (0-30 point scale) score on Day 29 compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jun Gu, MD, Principal Investigator — Suzhou Municipal Hospital
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No